CLINICAL TRIAL: NCT06182618
Title: Retrospective Analysis of Outpatient Intervention Effects in Patients With Metabolic Syndrome
Brief Title: Retrospective Analysis for Patients With Metabolic Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-1042
Record Dates: First submitted 2023-11-30; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-11

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Diet

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- low-carbohydrate diet: 20-30% carbohydrates, 40-45%fat, and 30-40%protein
  Interventions: Other: dietary, semaglutide or/and metformin
- balanced diet: 50-65% carbohydrate, 20-30% fat and 10-20% protein
  Interventions: Other: dietary, semaglutide or/and metformin
- pharmacotherapy: semaglutide (1mg per week) or/and metformin (o.5g three times a day)
  Interventions: Other: dietary, semaglutide or/and metformin

INTERVENTIONS:
Other: dietary, semaglutide or/and metformin — patients were prescribed dietary and pharmaceuticals for weight loss

SUMMARY:
The incidence of metabolic syndrome and related diseases is gradually increasing, and diet and medication are currently common outpatient treatment methods. This study retrospectively analyzes the clinical data of patients with metabolic syndrome and related diseases who have visited our outpatient department in the past 10 years, compares the therapeutic effects of different treatment methods on their blood glucose, blood lipids, blood pressure, uric acid, and body composition, and provides evidence support for clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

• individuals who had at least a 2 follow up visits with a BMI of 24 or more with the pri-mary goal of losing weight.

Exclusion Criteria:

* patients did not follow-up on a monthly basis;
* patients followed-up less than 1 times within 3 months;
* patients having incomplete data;
* patients changing their interventions during fol-low-ups

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This was a retrospective study of the weight loss effect in 1 to 3 months in overweight or obese individuals at the department of clinical nutrition in the Second Affiliated Hospital of Zhejiang University, School of Medicine in China between 1 January 2020 and 1 Janu-ary 2024.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
weight | 0month/1month/2months/3 months
  Weight was measured through multi-frequency bioelectrical impedance analysis InBody 720 (Bio Space Co., Seoul, Korea) at various time points

SECONDARY OUTCOMES:
visceral fat area(VFA) | 0month/1month/2months/3 months
  VFA was measured through multi-frequency bioelectrical impedance analysis InBody 720 (Bio Space Co., Seoul, Korea) at various time points
skeletal muscle mass(SMM) | 0month/1month/2months/3 months
  SMM was measured through multi-frequency bioelectrical impedance analysis InBody 720 (Bio Space Co., Seoul, Korea) at various time points

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China